CLINICAL TRIAL: NCT04999826
Title: Use of Multiscale Omics to Develop a Cohort Database and Study Platform in Breast Cancer Survivors
Brief Title: Multiscale Omics for the Development of a Cohort Database and Study Platform in Breast Cancer Survivors
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 19-005860; NCI-2021-07536 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-07-22; First posted 2021-08-11 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage 0 Breast Cancer AJCC v8; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage 0 Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, saliva, stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (questionnaire, biospecimen collection): Participants complete questionnaires over 10 minutes and undergo blood, urine, saliva, and fecal samples collection.
  Interventions: Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo biospecimen collection
  Other Names: Biological Sample Collection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study gathers information to create a database to improve the ability to diagnose cancer, predict long term health of breast cancer patients, and help develop future treatment products. This study will provide a foundational platform for therapeutic development and intervention studies in the future and may for therapeutic development and intervention studies in the future, and may advance researchers understanding of the contribution gut bacteria to altered circulating estrogens in breast cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To use multiscale omics to build a cohort database that can be used as a reference population in support of multivariate analysis, predictive modeling, and development of natural product therapeutics and precision medicine applications for breast cancer survivors.

SECONDARY OBJECTIVE:

I. To detect unique patterns of variance between 1) targeted serum metabolites, 2) plasma metabolome, 3) gut microbiome community structure, 4) gut microbiome metabolome, 5) urine metabolome, 6) quality of life measures, and 7) breast cancer survivors (BCS) symptoms by using multivariate analysis, machine learning tools, and artificial intelligence applied to the large data sets developed in this trial.

OUTLINE:

Participants complete questionnaires over 10 minutes and undergo blood, urine, saliva, and fecal samples collection.

ELIGIBILITY:
Inclusion Criteria:

* BCS GROUP
* Female patients diagnosed with breast cancer age 18 - 75, stages 0 through 3 at time of diagnosis
* Who have completed active therapy (including surgery, radiation, and/or chemotherapy)
* Able to speak English and complete surveys and provide the specimen (willing to follow the sample collection instructions)
* Able to read, understand and sign inform consent
* CONTROL GROUP
* Healthy Volunteers age 18 - 75
* Able to speak and read English, complete consent, surveys, and provide specimens

Exclusion Criteria:

* Unable to give written consent
* Unable to fast before providing blood and urine
* Pregnant women (per participant report) and males
* Unwilling to travel to Mayo Clinic Rochester to provide bio specimens

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer stages 0 through 3 at time of diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Utilization of multiscale omics to build a cohort database for breast cancer survivors | Up to 5 years

SECONDARY OUTCOMES:
Detection of unique patterns of variance | Up to 5 years
  Will be detected between 1) serum metabolites, 2) plasma metabolome, 3) gut microbiome community structure, 4) gut microbiome metabolome, 5) urine metabolome, 6) quality of life measures, and 7) BCS symptoms by using multivariate analysis applied to the large data sets developed in this trial.
Detection of unique patterns of variance | Up to 5 years
  Will be detected between 1) serum metabolites, 2) plasma metabolome, 3) gut microbiome community structure, 4) gut microbiome metabolome, 5) urine metabolome, 6) quality of life measures, and 7) BCS symptoms by using machine learning tools applied to the large data sets developed in this trial.
Detection of unique patterns of variance | Up to 5 years
  Will be detected between 1) serum metabolites, 2) plasma metabolome, 3) gut microbiome community structure, 4) gut microbiome metabolome, 5) urine metabolome, 6) quality of life measures, and 7) BCS symptoms by using artificial intelligence applied to the large data sets developed in this trial.

CONTACTS AND LOCATIONS:
Overall Officials: Brent A. Bauer, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials